CLINICAL TRIAL: NCT01403519
Title: Innovative Biomarkers in Alzheimer's Disease and Frontotemporal Dementia (FTD): Preventative and Personalized
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Prof' Judith Aharon-Peretz, Rambam Medical Center
Other Study IDs: 437-10CTIL
Record Dates: First submitted 2011-07-06; First posted 2011-07-27 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and CSF
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Alzheimer's disease patients: Patients blood and CSF samples
- Control group: Blood and CSF samples
- FTD patients: Blood ad CSF samples

SUMMARY:
Tau pathology and tangles have been associated with cognitive dysfunction causing neurodegeneration. AD, the most abundant tauopathy is characterized by amyloid plaques and tau tangles. An abundance of tau inclusions, in the absence of amyloid deposits, defines Pick's disease (frontotemporal lobar degeneration), progressive supranuclear palsy (PSP), corticobasal degeneration (CBD) and other diseases including frontal atrophy associated with cognitive clinical dysfunction of frontal dysexecutive syndrome, progressive nonfluent aphasia and semantic dementia as recently reviewed (Gozes 2010). It is the investigators aim to follow other protein expression [as per recent publications (Marksteiner et al., 2011)] in blood and CSF samples from those tauopathies.

Significance: Results should establish the possibility of using tau and other proteins as markers for early detection and disease progression in FTD, also in comparison to Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Assessing biomarkers in Alzheimer's disease and frontotemporal dementia

1. Specific Aims

   To enhance the field of biomarker recognition and facilitate preventative and personalized medicine we are now posing the following question, does the Israeli patient population present similar plasma protein profile as described before for other populations (Marksteiner et al., 2011).

   Studies will be carried out by RNA transcript quantification, quantitative real time polymerase chain reaction (blood cells and CSF) and immunochemical detection at the protein level (CSF and serum).
2. Methods:

Lymphocytes:

Human lymphocytes are isolated from 10 ml of venous blood using the Ficoll Paque method (de Rock and Taylor 1977; McCauley and Hartmann, 1982), for RNA extraction and determinations we shall follow-up the methods described in our manuscripts (Dresner et al., 2011).

Blood plasma and serum will be prepared as outlined in www.peoimmune.com. Protein quantitation will be carried out using the Tri reagent (Sigma) which allows for simultaneous preparation of RNA, DNA and protein and plasma immunodepletion and albumin depletion kits from Sigma.

Protein quantification: this will be carried out on cellular proteins and also on plasma proteins by SDS-polyacrylamide gel electrophoresis, followed by western analysis.

CSF samples will be collected through a spinal needle inserted into the L4-L5 or L3-L4 vertebral space with the subject in the lateral decubitus position. One ml of CSF derived from each patient will be immediately immersed in ice, with subsequent maintenance at -70 degrees C (or in dry ice during shipping) until the time of the assay. Half ml of each CSF sample will be concentrated by lyophilization in a Speed-Vac (Holten, Gydevang, Denmark) to about 0.1ml. CSF protein immunoblotting will be performed using a similar methodology as described above [and see also(Kozlovsky et al., 2004)]. Protein expression will be analyzed by western blots (Shiryaev et al., 2010).

Number of patients:

We estimate that about 30 patients with Alzheimer's disease, 20 patients with frontotemporal dementia and 20 controls will be included.

Professor Aharon-Peretz will evaluate patients with suspected Alzheimer's disease and frontotemporal dementia and include patients at various disease stages in a stratified manner (mild, moderate and severe). All patients will have signed an informed consent form, as per Helsinki guidelines. Clinical evaluation will include: physical and neurological evaluation. All patients will be asked to donate 50 ml blood and selected patients will undergo lumber puncture. The lumber puncture will be performed with the neurological work up. Professor Gozes will coordinate the scientific aspect of the study.

Study coordinators:

Scientific: Professor Illana Gozes, PhD, The Lily and Avraham Gildor Chair for the Investigation of Growth Factors; Director, The Adams Super Center for Brain Studies, Tel Aviv University: igozes@post.tau.ac.il Clinical material: Professor Judith Aharon-Peretz, MD, Head of "Cognitive Neurology Unit" Rambam Rambam-Health Care Campus, Haifa, Israel

ELIGIBILITY:
Inclusion Criteria:

* Minimal cognitive impairment (MCI) and Alzheimer's disease (AD) patients, men and women, age 45-80 will be asked to participate in the present study.
* MCI will be diagnosed when on cognitive evaluation the patients will score <1.5 SD on memory tests and will not be demented. AD will be diagnosed according to NINCDS-ADRDA research criteria. Patients will be stratified by age and cognitive (dementia) status. Disease severity for AD: mild to moderate (MMSE >16) AD.
* Frontotemporal dementia: patients with a clinical diagnosis of frontotemporal dementia [behavioral variants (bv)FTD, progressive nonfluent aphasia (PNFA), or semantic dementia] and the related syndromes corticobasal syndrome (CBS) and progressive supranuclear palsy (PSP) will be included.
* Inclusion criteria (controls): men and women, ages 45-80, willing to participate in the study and donate a blood samples.

Exclusion Criteria:

* (patients and controls):

  1. Subjects unable/unwilling to sign an informed consent.
  2. Patients with associated medical condition: alcoholism, immune diseases and end stage medical conditions.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We estimate that about 30 patients with Alzheimer's disease, 20 patients with frontotemporal dementia and 20 controls will be included.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Aharon-Peretz, M.D., Principal Investigator — Rambam Hospital, Haifa, Israel; Illana Gozes, Ph.D., Principal Investigator — Tel Aviv University, Sackler School of Medicine, Israel
Locations (1):
- Rambam Hospital, Haifa, Israel

REFERENCES:
- [Background] Gozes I. Tau pathology and future therapeutics. Curr Alzheimer Res. 2010 Dec;7(8):685-96. doi: 10.2174/156720510793611628. PMID 20678069
- [Background] Marksteiner J, Kemmler G, Weiss EM, Knaus G, Ullrich C, Mechtcheriakov S, Oberbauer H, Auffinger S, Hinterholzl J, Hinterhuber H, Humpel C. Five out of 16 plasma signaling proteins are enhanced in plasma of patients with mild cognitive impairment and Alzheimer's disease. Neurobiol Aging. 2011 Mar;32(3):539-40. doi: 10.1016/j.neurobiolaging.2009.03.011. Epub 2009 Apr 22. PMID 19395124
- [Background] de Rock E, Taylor N. An easy method of layering blood over Ficoll-Paque gradients. J Immunol Methods. 1977;17(3-4):373-4. doi: 10.1016/0022-1759(77)90120-x. No abstract available. PMID 562380
- [Background] McCauley I, Hartmann PE. The estimation of B lymphocytes and their subpopulations in pigs. A comparison between a method using whole blood and one using Ficoll-Paque purified mononuclear cells. J Immunol Methods. 1982;50(1):33-8. doi: 10.1016/0022-1759(82)90301-5. PMID 6979582
- [Background] Dresner E, Agam G, Gozes I. Activity-dependent neuroprotective protein (ADNP) expression level is correlated with the expression of the sister protein ADNP2: deregulation in schizophrenia. Eur Neuropsychopharmacol. 2011 May;21(5):355-61. doi: 10.1016/j.euroneuro.2010.06.004. Epub 2010 Jul 3. PMID 20598862
- [Background] Kozlovsky N, Regenold WT, Levine J, Rapoport A, Belmaker RH, Agam G. GSK-3beta in cerebrospinal fluid of schizophrenia patients. J Neural Transm (Vienna). 2004 Aug;111(8):1093-8. doi: 10.1007/s00702-003-0127-0. Epub 2004 Apr 27. PMID 15254796
- [Background] Shiryaev N, Jouroukhin Y, Gozes I. 3R tau expression modifies behavior in transgenic mice. J Neurosci Res. 2010 Sep;88(12):2727-35. doi: 10.1002/jnr.22431. PMID 20544828